CLINICAL TRIAL: NCT01884285
Title: A Phase I, Open-label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Anti-tumour Activity of AZD8186 in Patients With Advanced Castration-resistant Prostate Cancer (CRPC), Squamous Non-Small Cell Lung Cancer (sqNSCLC), Triple Negative Breast Cancer (TNBC) and Patients With Known PTEN-deficient/Mutated or PIK3CB Mutated/ Amplified Advanced Solid Malignancies as Monotherapy and in Combination With Abiraterone Acetate or AZD2014
Brief Title: AZD8186 First Time In Patient Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4620C00001
Record Dates: First submitted 2013-06-17; First posted 2013-06-24 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Advanced Castrate-resistant Prostate Cancer CRPC; Squamous Non-Small Cell Lung Cancer sqNSCLC; Triple Negative Breast Cancer TNBC
Keywords: Advanced Castrate-resistant Prostate Cancer(CRPC); Squamous Non-Small Cell Lung Cancer(sqNSCLC); Triple Negative Breast Cancer(TNBC); PTEN-deficient/mutated Advanced Solid Malignancies; PIK3CB mutated/amplified advanced solid malignancies
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — AZD8186

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: AZD8186 monotherapy (Experimental): Patients will receive a single dose on Day 1 followed by ongoing multiple dosing. The initial schedule will use intermittent dosing of AZD8186.
  Interventions: Drug: Part A: AZD8186 monotherapy
- Part C2: AZD8186/abiraterone (Experimental): Patients will receive a week of abiraterone acetate with prednisone followed by combination dosing with AZD8186.
  Interventions: Drug: Part C2: Abiraterone acetate combination with AZD8186
- Part D1: AZD8186 and AZD2014 (Experimental): Combination dosing with AZD8186 and AZD2014 both given on an intermittent schedule at escalating dose levels of each IMP for combination dose finding
  Interventions: Drug: Part D1: AZD2014 combination with AZD8186
- Part B: AZD8186 monotherapy (Experimental): Part B - multiple dosing of intermittent dose schedule
  Interventions: Drug: Part B: AZD8186 monotherapy
- Part D2: AZD8186/ AZD2014 (Experimental): Expanded cohort of patients will be treated at a tolerated combination dose level established in Part D1
  Interventions: Drug: Part D2 AZD2014 combination with AZD8186
- Part C1: AZD8186 & abiraterone (Experimental): Patients will receive a week of abiraterone acetate with prednisone followed by combination dosing with AZD8186 at escalating doses of AZD8186 for the purpose of dose finding
  Interventions: Drug: Part C1: Abiraterone acetate combination with AZD8186

INTERVENTIONS:
Drug: Part A: AZD8186 monotherapy — The initial schedule will use intermittent dosing of AZD8186. Dose, frequency and schedule in subsequent cohorts may be modified in response to safety, tolerability, pharmacokinetic and preclinical data.
  Arms: Part A: AZD8186 monotherapy
Drug: Part B: AZD8186 monotherapy — Part B will be at a dose(s) and schedule(s) at or below from Part A
  Arms: Part B: AZD8186 monotherapy
Drug: Part C1: Abiraterone acetate combination with AZD8186 — Dose and schedule finding of AZD8186 added to approved labelled dose of abiraterone acetate (with prednisone).
  Arms: Part C1: AZD8186 & abiraterone
Drug: Part D1: AZD2014 combination with AZD8186 — Dose & schedule finding of AZD8186 in combination with AZD2014
  Arms: Part D1: AZD8186 and AZD2014
Drug: Part D2 AZD2014 combination with AZD8186 — Combination AZD8186/ AZD2014 dose expansion at dose determined in Part D1
  Arms: Part D2: AZD8186/ AZD2014
Drug: Part C2: Abiraterone acetate combination with AZD8186 — Dose expansion of AZD8186 at dose determined in Part C1 added to approved dose of abiraterone acetate (with prednisone)
  Arms: Part C2: AZD8186/abiraterone

SUMMARY:
This is a phase I, open-label, multicentre study of AZD8186 administered orally in patients with advanced castrate-resistant prostate cancer (CRPC), squamous non-small cell lung cancer (sqNSCLC), triple negative breast cancer (TNBC) and known PTEN-deficient/mutated or PIK3CB mutated/amplified advanced solid malignancies as monotherapy and in combination with abiraterone acetate or AZD2014.

DETAILED DESCRIPTION:
This is a phase I, open-label, multicentre study of AZD8186 administered orally in patients with advanced castrate-resistant prostate cancer (CRPC), squamous non-small cell lung cancer (sqNSCLC), triple negative breast cancer (TNBC) and known PTEN-deficient/mutated or PIK3CB mutated/amplified advanced solid malignancies. The study design allows an escalation of dose with intensive safety monitoring to ensure the safety of the patients.

There are 4 parts to this study: Part A, monotherapy dose escalation, Part B, monotherapy expansion cohort(s) in PTEN deficient patients at the monotherapy intended therapeutic dose(s) and schedule(s), Part C, AZD8186 added to abiraterone accetate (with prednisone) treatment - dose/ schedule finding followed by expansion phase in PTEN-deficient/mutated or PIK3CB mutated mCRPC and Part D, AZD8186 in combination with AZD2014 (a novel dual mTORC1/2 inibitor) dose/schedule finding followed by expansion phase in PTEN-deficient/mutated or PIK3CB mutated TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Male or female, aged 18 years and older
* Histologically or cytologically proven diagnosis of prostate cancer, sqNSCLC, TNBC, or known PTEN-deficient solid malignancy, and is refractory to standard therapies.
* Females should be using adequate contraceptive measures, not be breast feeding and must have negative pregnancy test prior to start of dosing if of child-bearing potential
* WHO/ECOG performance status 0 to 1 with no deterioration over the previous 2 weeks and min life expectancy of 12 weeks
* Tumours that are known to have genomic alterations in PTEN or PIK3CB by local test results may also be eligible.

Part B - Tumour amenable to taking of paired biopsies in opinion of the investigator.Patients with TNBC or mCRPC: PTEN-deficient tumours

Parts A,B or D1(mCRPC)

* PSA at screening must be ≥2 µg/L.
* Preceding line of treatment included response to anti-androgen, progression documented after withdrawal of the anti-androgen.
* Serum testosterone concentration ≤50 ng/dL sustained by medical or surgical castration

Parts A,B or D (TNBC)

- Oestrogen receptor, progesterone receptor and HER2 negative advanced adenocarcinoma of breast.

Parts A, B or D1 (solid malignancies) - Consented provision of formalin fixed paraffin embedded blocks/ slides from most recent tissue sample.

Part C (all patients):

* May have received treatment with abiraterone acetate, enzalutamide and/or one prior chemotherapy (docetaxel)
* Serum testosterone concentration ≤50 ng/dL sustained by medical or surgical castration.
* Early or confirmed evidence of progressive disease.
* Last PSA value should have increase of ≥ 25% of the first PSA value and an absolute increase of ≥2 ng/mL over the first PSA value
* Serum potassium > 3.5 mmol/L

Parts C2 and D2

- Prospectively determined eligible PTEN alteration determined by next generation sequencing, protein deficient determined by IHC or PIK3CB mutation/amplification.

Part D2

- Measurable disease (at least 1 lesion ≥10 mm longest diameter or for lymph nodes short axis ≥15 mm) by CT/MRI

Exclusion Criteria

* Treatment before study with

  1. Nitrosourea or mitomycin C within 6 weeks
  2. Investigational agents from previous clinical study within 4 weeks
  3. Chemotherapy, immunotherapy or anticancer agents within 4 weeks
  4. hormonal therapy
* Treatment before study with

  1. Strong inhibitors and strong or moderate inducers of CYP3A4
  2. Radiotherapy with a wide field of radiation within 4 weeks,
* With the exception of alopecia or toxicities related to the use of gonadotropin-releasing hormone agonists any unresolved toxicities from prior therapy greater than CTCAE grade 1 at time of study treatment
* Spinal cord compression or brain metastases unless asymptomatic treated and stable and not requiring steroids
* Evidence of severe or uncontrolled systemic diseases including active liver disease (other than malignancy), active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).

Exclusion crtieria Part C

* Pre-existing Grade 2 or higher chronic diarrhoea
* Major bowel surgery which in the opinion of the Investigator should exclude the patient
* Use of antibiotics to treat chronic infections within 28 days prior to first dose
* Sensitive or narrow therapeutic range substrates of CYP2D6
* Severe or moderate hepatic impairment
* Persistent uncontrolled hypertension (systolic >160 mmHg/ diastolic >100 mmHg

Exclusion Criteria Part D

* Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 and CYP2C8 if taken within the stated washout periods before the first dose
* Exposure to sensitive or narrow therapeutic range substrates of the drug metabolising enzymes CYP2C8, CYP2C9, CYP2C19 or the drug transporters Pgp, BCRP, OATP1B1, OATP1B3, OCT1 and OCT2 within the appropriate wash-out period before the first dose of study treatment.
* Haemopoietic growth factors within 2 weeks prior to receiving study drug.
* Patients who have experienced any of the following procedures or conditions currently or in the preceding 12 months: coronary artery bypass graft, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association Grade ≥2, supraventricular arrhythmias including atrial fibrillation, which are uncontrolled, haemorrhagic or thrombotic stroke, including transient ischaemic attacks or any other central nervous system bleeding.
* Abnormal ECHO or MUGA at baseline <55%.
* Patients with Diabetes Type I or uncontrolled Type II as judged by the Investigator

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Routine safety assessments, throughout the period that patients receive AZD8186 up to 30 days following discont of last dose of study treatment.
  Assess safety and tolerability of AZD8186 when given as monotherapy or in combination with abiraterone acetate (with prednisone) or with AZD2014 by measuring AEs, SAE (incl death), safety measures incl ECG, physical exam, pulse, blood pressure, weight, lab variables

SECONDARY OUTCOMES:
Part A: The number of evaluable patients with dose limiting toxicities (DLTs). | DLTs assessed during the first 21 days of multiple dosing.
  Measure the number of evaluable patients with reported dose limiting toxicities (DLTs) at escalating dose levels and different intermittent and continuous dose schedules of AZD8186 monotherapy
Part A, B, C + D: Antitumor activity of AZD8186 monotherapy or in combination | Every 12 weeks (non prostate patients) or every 6 weeks (prostate patients) from baseline up to disease progression or withdrawal of consent
  Evaluation of tumour response using RECIST 1.1 or Prostate Cancer Clinical Trials Working Group (PCWG2) criteria for those patients with prostate cancer
Part A, B, C and D: Anti-tumour activity of AZD8186 monotherapy or in combination | PSA at Screening, Days 1, 8 & 15 then every 28 days, discontinuation of treatment (on average after 4 months), 30-day follow-up: CTC enumeration Days 1, 56 & 84, then every 12 weeks, at discontinuation (on average after 4 months).
  Measurement of changes in circulating prostate-specific antigen (PSA) and circulating tumour cells (CTC) enumeration in pts with prostate cancer.
Part A + B: Plasma concentrations of AZD8186 and pharmacokinetic parameters (Cmax, tmax, AUC, terminal rate constant, clearance, half life, volume of distribution and mean resistance time) | Prior to first dose and during first 28 days of treatment
  Blood samples will be collected at multiple timepoints on 2 intense PK collection days, with sparse sampling on additional days.
Part A + B: 4 beta-hydroxy cholesterol concentration in blood samples. | Blood samples will be collected from all patients for 4 beta-hydroxy cholesterol concentration measurements pre-dose day 1 and pre-morning dose day 22 in both Part A and B.
  Understanding of the CYP3A4 induction potential of AZD8186
Part B: Obtaining a preliminary assessment of the antitumour activity of AZD8186 as monotherapy | Paired tumour biopsies will be collected; one prior to treatment and the other during treatment (after at least 3 consecutive days of dosing 2-4 hours post-dose during 2nd week of trreatment)
  Evaluation of proof of mechanism biomarkers in PTEN-deficient TNBC or mCRPC tumour tissue
Part B: Obtaining a preliminary assessment of AZD8186 drug effect in the tumour | Paired tumour biopsies will be collected; one prior to treatment and the other during treatment (after at leat 3 consecutive days of dosing 2-4 hours post-dose in the second week of treatment)
  Evaluation of pharmacodynamics biomarker changes in tumour tissue
Part A: Urine concentrations of AZD8186 and pharmacokinetic parameters (Cmax, tmax, AUC, terminal rate constant, clearance, half life, volume of distribution and mean residence time) | Urine samples will collected at multiple time points: Day 1 (predose, 15min post dose, 30min post dose); Last dosing day during week 3 (predose and 15min post dose)
  Evaluation of the pharmacokinetics of AZD8186
Part C: safety and tolerability assessed by dose limiting toxicity of AZD8186 with abiraterone acetate (and prednisone) | DLTs assessed during the first 21 days of multiple dosing
  Dose limiting toxicity of AZD8186 when given at different doses and schedules in combination with abiraterone (with prednisone)
Part C: pharmacokinetics of and exposure to AZD8186, its major metabolite M1, and abiraterone | Blood samples will be collected at multiple timepoints on 2 intense PK collection days between screening and the end of the first 28 days of combination treatment.
  Assess the impact of co-administration on pharmacokinetics of and exposure to AZD8186, its major metabolite M1, and abiraterone
Part C: steady state exposure to abiraterone | Blood samples will be collected at multiple timepoints on 2 intense PK collection days between screening and the end of the first 28 days of combination treatment.
  Measure the steady state exposure to abiraterone in the absence and presence of steady state AZD8186
Part C: steady state exposure of AZD8186 in combination with abiraterone acetate | Blood samples will be collected at multiple timepoints on 2 intense PK collection days between screening and the end of the first 28 days of combination treatment.
  Measure the steady state exposure of AZD8186 in combination with abiraterone acetate and compare to previous steady state exposures when administered as a monotherapy
Part D: Measure the dose limiting toxicity of AZD8186 in combination with AZD2014. | DLTs assessed during the first 21 days of multiple dosing
  Safety and tolerability of the combination of AZD8186 and AZD2014
Part D: Single dose and multiple dose pharmacokinetics of and assess exposure to AZD8186, its major metabolite M1, and AZD2014 when co-administered | Blood samples will be collected at multiple timepoints on intense PK collection days for AZD8186 and AZD2014 monotherapy run-in, cycle 0 (single dose), day 9 (multiple dose)
  Measure the pharmacokinetics of and exposure to AZD8186, its major metabolite M1, and AZD2014 when co-administered
Part D: Measure the exposure to AZD2014 following the last weekly dose of AZD2014 in the absence and presence of multiple dose AZD8186. | Blood samples will be collected at multiple timepoints on intense PK collection days for AZD8186 and AZD2014 monotherapy run-in, cycle 0 (single dose), Day 9 of treatment (multiple dose)
  Assessment of exposure to AZD2014 in absence and presence of multiple dose AZD8186
Part D: Measure the exposure on the 4th administred dose of AZD8186 in the absence and presence of multiple dose AZD2014 | Blood samples will be collected at multiple timepoints on intense PK collection days for AZD8186 and AZD2014 monotherapy run-in, cycle 0 (single dose), day 9 (multiple dose)
  Assessment of exposure of AZD8186 in absence and presence of multiple dose AZD2014

CONTACTS AND LOCATIONS:
Overall Officials: Michele Mochetta, MD, Study Director — AstraZeneca; Lillian Siu, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (12):
- United States (5):
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Research Site, Toronto, Ontario, Canada
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Pozuelo de Alarcón
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home